CLINICAL TRIAL: NCT00623402
Title: Combined Treatment of Sorafenib and Pegylated Interferon α2b in Stage IV Metastatic Melanoma: a Prospective Non-randomized, Multicenter Phase II Study
Brief Title: Combined Treatment of Sorafenib and Pegylated Interferon α2b in Stage IV Metastatic Melanoma
Acronym: SoraPeg
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital Schleswig-Holstein (Other)
Collaborators: Dermatologic Cooperative Oncology Group (Other)
Responsible Party: Axel Hauschild, MD, University Hospital Schleswig-Holstein
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DeCOG SoraPeg 2007; EudraCT 2007-001918-16
Record Dates: First submitted 2008-02-01; First posted 2008-02-26 (Estimated); Last update posted 2011-01-12 (Estimated); Status verified 2008-02

CONDITIONS: Melanoma
Keywords: Metastatic melanoma; Pegylated interferon; Protein Kinase Inhibitors; Sorafenib; PegIntron; Therapeutic Uses; melanoma (skin)
MeSH Terms: conditions — Melanoma | interventions — Sorafenib; peginterferon alfa-2b

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- A (Experimental)
  Interventions: Drug: Sorafenib; Drug: pegylated interferon α-2b

INTERVENTIONS:
Drug: Sorafenib — 2x 400 mg orally per day (4 tablets)
Drug: pegylated interferon α-2b — 3 µg/kg body weight s.c. once a week
  Other Names: PegIntron

SUMMARY:
To evaluate the efficacy and safety of a combined treatment with Sorafenib (Nexavar®) and pegylated interferon-α-2b (PegIntron®) in patients with malignant melanoma in stage IV.

DETAILED DESCRIPTION:
This is a a prospective non-randomized, multicenter Phase II Study to evaluate the efficacy and safety of a combined treatment with Sorafenib (Nexavar®) and pegylated interferon-α-2b (PegIntron®) in patients with malignant melanoma in stage IV.

The investigators will determine disease control rate (CR,PR,SD) after 8 weeks of treatment with pegylated interferon- α-2b (3 µg/kg body weight s.c. once a week) combined with Sorafenib 2x 400 mg (2 tablets orally, twice daily)

ELIGIBILITY:
Inclusion Criteria:

* Histologically documented metastatic melanoma classified as stage IV (AJCC 2002) of cutaneous origin.
* ≥ 18 years of age
* ECOG performance status of 0 or 1
* Patients should not have received any systemic treatment for stage IV disease (study = "first-line" treatment).
* Patients with progressive disease (PD) to stage IV under prior treatment with interferons as well as all patients who have already been treated with Sorafenib should not be included.

The following are allowed:

* adjuvant interferon treatment (without progressive disease during treatment!) or vaccine therapy for resected stage I-III disease
* palliative surgery or radiotherapy for stage IV disease
* prior cytokine or chemotherapy treatment for local-regional disease by isolated limb perfusion or intralesional therapy
* Life expectancy >6 months.
* Patients must have measurable disease defined as >= 1 not pretreated unidimensional measurable lesion >= 20 mm (conventional techniques) or >= 10 mm by spiral CT/MRI.

Patients must have adequate hematological, renal and liver functions as defined by laboratory values below performed within 14 days prior to study inclusion:

* absolute neutrophil count (ANC) > 1.5 x 109/l
* platelet count > 100 x 109/l
* hemoglobin > 10 g/dl (> 6.2 mmol/l)
* serum creatinine <= 1.5 x upper limit of institutional values
* total serum bilirubin <= 1.5x upper limit of institutional values
* ALAT and ASAT <= 2.5x upper limit of institutional values (exception: liver metastases)

In addition:

* Patients should not suffer from frequent vomiting or medical conditions which could interfere with oral medication intake.
* Negative pregnancy test of women of childbearing potential performed within 7 days prior to the start of treatment.
* Women of childbearing potential must agree to use an effective method of contraception (Pearl-Index < 1, e.g. hormonal contraception including the combined oral contraceptive pill, the transdermal patch, and the contraceptive vaginal ring, intrauterine devices or sterilization) during treatment and for at least 6 months thereafter.
* Men must agree to use an effective method of contraception during treatment and for at least 6 months thereafter.
* Patients should understand the informed consent and will need to sign the consent

Exclusion Criteria:

* Ocular or mucosal melanoma.
* History or evidence of brain metastasis.
* Patients with LDH values higher than 2x upper limit of institutional values.
* Patients with thyroid dysfunctions not responsive to therapy.
* Patients with uncontrolled diabetes mellitus.
* Patients with prior or active autoimmune disease or autoimmune hepatitis.
* Cardiac disease: congestive heart failure > class II NYHA, patients must not have unstable angina or new onset of angina or myocardial infarction within the past 6 months. Cardiac ventricular arrhythmias requiring antiarrhythmic therapy.
* Uncontrolled hypertension defined as systolic blood pressure > 150 mm Hg or diastolic pressure > 90 mm Hg, despite optimal management.
* Active clinically serious infections > CTCAE Grade 2.
* Patients who are HIV positive or have AIDS.
* Thrombotic or embolic events including transient ischemic attacks within the past 6 months.
* Evidence or history of bleeding diathesis or coagulopathy.
* Therapeutic anticoagulation with Vitamin K antagonists such as warfarin, or with heparins or heparinoids. Low dose warfarin is permitted if INR is < 1.5. Low dose aspirin is permitted.
* Known or suspected allergy to Sorafenib or any ingredient of Sorafenib or PEG-IFN-α -2b or any ingredient of PEG-IFN-α -2b or to any interferone.
* Previous cancer that is distinct in primary site or histology from melanoma except cervical cancer in situ, treated basal cell carcinoma, superficial bladder tumors or any cancer curatively treated 3 years prior to study entry.
* Substance abuse, medical or psychological condition that may interfere with the patient´s participation in the study.
* Patients with medication requiring chronic systemic corticosteroids.
* Patients with prior systemic anticancer treatment in the last 2 weeks.
* Patients with severe liver disease or severe renal disease.
* Patients with seizure disorders requiring anticonvulsant therapy.
* Patients with any severe debilitating diseases.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Estimated)
Dates: Start 2008-01; Primary Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
disease control rate (CR,PR,SD) | 8 week staging

SECONDARY OUTCOMES:
Best response | 12 months
Progression free survival (PFS) | During active treatment
Overall survival | 48 week follow-up
Safety and tolerability of the combined treatment | During active treatment

CONTACTS AND LOCATIONS:
Overall Officials: Axel Hauschild, MD, Study Director — UK-SH Department of Dermatology
Locations (10):
- Germany (10):
  - Dpt. of Dermatology, Humboldt University, Berlin
  - Dept. of Dermatology, Elbe Klinikum, Buxtehude
  - Dpt. of Dermatology, University of Cologne, Cologne
  - Dpt. of Dermatology, University of Hannover, Hanover
  - Dpt. of Dermatology, University of Homburg/Saar, Homburg/Saar
  - Dpt. of Dermatology; UK-SH Campus Kiel, Germany, Kiel
  - Dpt. of Dermatology, University of Mannheim, Mannheim
  - Dpt. of Dermatology, Ludwig-Maximilian-University, München
  - Dpt. of Dermatology, University of Tübingen, Tübingen
  - Dpt. of Dermatology, University of Würzburg, Würzburg

REFERENCES:
- See also: Official website of the Dermatologic Cooperative Oncology Group — http://www.ado-homepage.de